CLINICAL TRIAL: NCT02308813
Title: Predictability of Braking Performance in Patients With Degenerative Disease of the Hip Joint or With Total Hip Arthroplasty
Brief Title: Predictability of the Ability to Perform an Emergency Stop With Disorders of the Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 503/2014BO2
Record Dates: First submitted 2014-10-27; First posted 2014-12-04 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2014-11

CONDITIONS: Osteoarthritis; Total Hip Arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Braking and functionality with hip osteoarthritis (Experimental): Cohort testing of driving performance in a drive simulator and correlation with clinical functionality in patients with hip osteoarthritis
  Interventions: Other: Braking and functionality
- Braking and functionality with hip arthroplasty (Experimental): Cohort testing of driving performance in a drive simulator and correlation with clinical functionality in patients with total hip arthroplasty
  Interventions: Other: Braking and functionality

INTERVENTIONS:
Other: Braking and functionality

SUMMARY:
Several studies exist on patient performance in drive simulators especially around and after surgery. Recommendations concerning the ability to drive preoperatively are based on these studies, which generated their data using drive simulators. However, in all the datasets driving performance remains highly individual. Since a drive simulator is not readily available in normal general practitioner surgeries it would be helpful to have convenient clinical tests to evaluate a patients individual ability to perform an emergency stop. This study aims at evaluating different possibilities how such performance might be predicted. Patients with hip osteoarthritis and patients who have received total hip arthroplasty are tested clinically and their results are compared with the gold standard experiment - a drive simulator.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 y
* valid driving license
* male and female
* Hip Osteoarthritis, Total hip arthroplasty
* capability to walk with or without a walking stick

Exclusion Criteria:

* myocardial infarction/Apoplexia < 6 months
* Total hip arthroplasty <5 weeks
* New York Heart Association 3/4
* lacking drivers' license
* peripheric sensomotor deficit <3/5 British Medical Research Council
* new fracture of the lower extremity or spine
* systemic or metastasised Cancer
* drug intake with centrally acting substances known to affect reaction time (Opioids, e.g. Tramadol, oxycodone, morphine, Til

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Correlation of an index of manual reaction time combined with functional hip tests and braking performance | Osteoarthritis group: cross sectional at consultation, Total hip arthroplasty group: cross-sectional - from 5 weeks postoperatively until 400 months postoperatively, at consultation
  Evaluation of degree of correlation of braking performance (total brake response time) and clinical testing of hip functionality in patients with hip osteoarthritis or total hip arthroplasty. The measure is a composite measure of multiple different tests. If a sufficient correlation between the composite measure and braking performance is observed a regression model will be developed.
  One time point of evaluation for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf K Hofmann, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Department of Orthopaedics, Tübingen, Germany

REFERENCES:
- [Background] Hau R, Csongvay S, Bartlett J. Driving reaction time after right knee arthroscopy. Knee Surg Sports Traumatol Arthrosc. 2000;8(2):89-92. doi: 10.1007/s001670050192. PMID 10795670